CLINICAL TRIAL: NCT02329184
Title: Safety, Tolerability, Preliminary Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of MYK-461 in Patient Volunteers With Hypertrophic Cardiomyopathy
Brief Title: Study Evaluating the Safety, Tolerability and Preliminary Pharmacokinetics and Pharmacodynamics of MYK-461
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MyoKardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYK-461-001
Record Dates: First submitted 2014-12-19; First posted 2014-12-31 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MYK-461 (Experimental)
  Interventions: Drug: MYK-461

INTERVENTIONS:
Drug: MYK-461

SUMMARY:
The purpose of this study is to establish initial safety, tolerability, pharmacokinetics and pharmacodynamics of MYK-461 in human subjects. This is a sequential group, single ascending (oral) dose study in NYHA Class I, II, or III patient volunteers aged 18-65 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCM
* Normal left ventricular ejection fraction (LVEF)
* NYHA class I, II or III

Exclusion Criteria:

* Inherited metabolic disorders, myocardial infiltration or cardiofaciocutaneous syndrome (e.g., Noonan's, Fabry's).
* History of clinically important atrial or ventricular arrhythmias
* History of positive human immunodeficiency virus (HIV) test and/or seropositive for hepatitis C virus (HCV) or hepatitis B virus (HBV)..

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 28 Days

SECONDARY OUTCOMES:
Determination of pharmacokinetics parameters as measured by Cmax | 28 Days
  maximum concentration (Cmax)
Determination of pharmacokinetics parameters as measured by Tmax | 28 Days
  time of the maximum measured concentration (Tmax)
Determination of pharmacokinetics parameters as measured by AUC | 28 Days
  area under the concentration-time curve (AUC)
Determination of pharmacokinetics parameters as measured by t1/2 | 28 Days
  half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Fox, MD, PhD, Study Director — MyoKardia, Inc.
Locations (7):
- United States (7):
  - Scottsdale, Arizona
  - Cypress, California
  - Stanford, California
  - Boston, Massachusetts
  - Kalamazoo, Michigan
  - Durham, North Carolina
  - Nashville, Tennessee